CLINICAL TRIAL: NCT07167420
Title: RISE Ileocecal Valve Functional Reconstruction for the Prevention of Postoperative Intestinal Dysfunction After Robotic/Laparoscopic Right Hemicolectomy: a Single-blind, Two-arm, Multicenter Randomized Controlled Clinical Study
Brief Title: RISE Ileocecal Valve Functional Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Army Medical University, China (Other)
Responsible Party: Principal Investigator, Weidong Xiao, Chief of General Surgery, Army Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RISE anastomosis 002
Record Dates: First submitted 2025-09-01; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Right-sided Colon Cancer
Keywords: right-sided colon cancer; laparoscopic surgery; ileocecal valve

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISE anastomosis (Experimental): After performing a conventional right hemicolectomy, an additional step is carried out in which sutures are used to artificially reconstruct an ileocecal valve structure at the ileal stump before proceeding with the ileocolic anastomosis.
  Interventions: Procedure: RISE (Revolute Insert Side-End ileocecal valve reconstruction)
- Control (No Intervention): Conventional right hemicolectomy was performed, with the ileocecal valve included in the resection.

INTERVENTIONS:
Procedure: RISE (Revolute Insert Side-End ileocecal valve reconstruction) — After performing a conventional right hemicolectomy, an additional step is carried out in which sutures are used to artificially reconstruct an ileocecal valve structure at the ileal stump before proceeding with the ileocolic anastomosis.
  Arms: RISE anastomosis

SUMMARY:
The traditional surgical treatment for right-sided colon cancer involves the removal of an important structure, the ileocecal valve, which includes the ileocecal valve. This can lead to problems such as diarrhea and malnutrition in patients. This study reconstructs an artificial ileocecal valve through intraoperative suturing to compensate for the function of the original ileocecal valve. The control group will undergo the routine resection of the right-sided colon, including the ileocecal valve. This is a randomized controlled study. Patients enrolled will be randomly assigned to the experimental group (ileocecal valve reconstruction during surgery) or the control group (no ileocecal valve reconstruction), with no differences in other treatment procedures. After a series of follow-up observations, the research team will analyze the safety and effectiveness of the method of ileocecal valve reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-80 years;
* ASA score ≤ 3;
* Patients newly diagnosed with tumors located in the appendix, ileocecal region, ascending colon, hepatic flexure of the colon, or the right one-third of the transverse colon, or those scheduled to undergo laparoscopic radical right hemicolectomy;
* No history of other gastrointestinal diseases (except for intestinal polyps or gallstones);
* Willing to participate in the study and sign the informed consent form;
* Complete clinical data available.

Exclusion Criteria:

* Presence of other malignant tumors in different organs;
* Tumor invasion into adjacent organs;
* Patients with concurrent infectious diseases or autoimmune diseases (e.g., Crohn's disease);
* Patients with congenital or acquired metabolic disorders;
* Use of antibiotics or other microbiota-altering medications within one month prior to enrollment;
* Changes in surgical plan resulting in the resection not including the ileocecal valve.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to first formed stool after surgery (Bristol stool score < 4). | 1 week after surgery
  According to the Bristol stool scale, stools are categorized into seven types. Since stool form is related to the duration of colonic transit, the scale can be used to assess intestinal transit time and evaluate anastomotic function. A score >5 is defined as diarrhea, with a score of 6 indicating mild diarrhea and a score of 7 indicating severe diarrhea.

SECONDARY OUTCOMES:
Operation time | during the surgery
anastomosis time | during surgery
intraoperative blood loss | during surgery
Complications within 30 days after surgery | 30 days after surgery
  Surgical complications evaluation was based on the Clavien-Dindo complication scoring system.
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusionsand total parenteral nutritionare also included. Grade III Requiring surgical, endoscopic or radiological intervention Grade IV Life-threatening complication (including CNS complications)* requiring IC/ICU-management Grade V Death of a patient
anastomosis healing | 3 months, 6 months and 1 year after surgery
  Colonoscopy is used to assess the healing status of an anastomosis, and to determine whether stenosis, ulcers, or other pathological changes have occurred.
albumin level | 3 days, 1 month, 3 months, 6 months and 1 year after surgery.
  for assessing the nutritional status.
bile acid | 3 days, 1 month, 3 months, 6 months and 1 year after surgery
  for assessing the nutritional status.
VitB12 | 3 days, 1 month, 3 months, 6 months and 1 year after surgery
  for assessing the nutritional status.
total protein | 3 days, 1 month, 3 months, 6 months and 1 year after surgery
  for assessing the nutritional status
EORTCQLQ-C30 | baseline, 1 month after surgery.
  for assessing quality of life after surgery
EORTCQLQ-CR2930 | baseline, 1 month after surgery.
  for assessing quality of life after surgery
gut microbiota | 1 month, 3 months, 6 months and 1 year after surgery.
  Analyzing the changes in gut microbiota through the patient's fecal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Xiao, MD, Principal Investigator — Department of General Surgery, Xinqiao Hospital, Army Medical University, No.183 Xinqiao Road, Chongqing, 400037, China

IPD SHARING:
Plan to Share IPD: No
After the completion of this study, the data will be made public and anyone can request it by email.

DOCUMENTS (2):
  • Study Protocol (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT07167420/Prot_000.pdf
  • Informed Consent Form (2025-07-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT07167420/ICF_001.pdf